CLINICAL TRIAL: NCT06663176
Title: Phase 1/2a Trial to Evaluate the Safety, Tolerability and Efficacy of Nebulised RESP30X Nitric Oxide Formulations in Non-Cystic Fibrosis Bronchiectasis (NCFB) Patients with Pseudomonas Aeruginosa (Pa) or Other Potentially Pathogenic Micro-organisms (PPMs)
Brief Title: Nebulised RESP30X Nitric Oxide Formulations in NCFB Patients with Pseudomonas Aeruginosa (Pa)
Acronym: NOPA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Thirty Respiratory Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RESP30X-001
Record Dates: First submitted 2024-10-25; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Non-Cystic Fibrosis Bronchiectasis
Keywords: Nitric Oxide

STUDY DESIGN:
Intervention Model Description: Single Ascending Dose, Multiple Daily Dosing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part 1-1 (Active) (Experimental): RESP303 Single Ascending Dose Phase followed by Multiple Daily Dosing (28-days)
  Interventions: Drug: RESP303
- Part 2-1 (Active) (Experimental): RESP302 TID Single Ascending Dose Phase followed by Multiple Daily Dosing (28-days)
  Interventions: Drug: RESP302
- Part 2-2 (Active) (Experimental): RESP303 BID Single Ascending Dose Phase followed by Multiple Daily Dosing (28-days)
  Interventions: Drug: RESP303
- Part 2-3 (Active) (Experimental): RESP303 TID Single Ascending Dose Phase followed by Multiple Daily Dosing (28-days)
  Interventions: Drug: RESP303

INTERVENTIONS:
Drug: RESP302 — Nitric Oxide agent
  Arms: Part 2-1 (Active)
Drug: RESP303 — Nitric Oxide agent
  Arms: Part 1-1 (Active); Part 2-2 (Active); Part 2-3 (Active)

SUMMARY:
A Phase 1/2a, Multi-Centre, Randomised, Open-label study to assess the safety, tolerability, PK, and efficacy of RESP30X in Adult NCFB participants with confirmed high-titre respiratory PPMs.

DETAILED DESCRIPTION:
A total of approximately 60 participants will be enrolled in this study, to give 30 participants completing the study.

Part 1: Approximately 12 NCFB patients with confirmed high-titre Pa (≥10^5 CFU/mL) to be enrolled to give 6 participants completing the study.

Participants will receive treatment with nebulised RESP303 in a Single Ascending Dose (SAD) phase followed by RESP303 three times a day (TID) multiple daily dosing for 28-days.

A safety review committee will meet after 6 participants have completed the study to determine whether Part 2 of the study can be initiated.

Part 2: Approximately 48 NCFB patients with confirmed high-titre respiratory PPMs (≥10^5 CFU/mL) to be enrolled to give 24 participants completing the study.

Participants will be randomised to receive treatment with nebulised RESP302 in a SAD phase, followed by RESP302 TID multiple daily dosing for 28-days, or nebulised RESP303 in a SAD phase, followed by either RESP303 twice a day (BID) or RESP303 TID multiple daily dosing for 28-days (1:1:1).

ELIGIBILITY:
Inclusion Criteria:

* Provide written, informed consent prior to all study-related procedures and agree to undergo all study procedures.
* Aged between 18 and 75 years, inclusive.
* Clinical history of bronchiectasis affecting 1 or more lobes based on symptoms (cough, sputum productive and/or recurrent lower respiratory tract infections) as confirmed by historical CT scan and radiology report performed within the last 5 years.
* Confirmed high-titre respiratory PPMs (Part 1: Pa only) at screening ≥10^5 CFU/mL (as determined by central laboratory microbiological cultures).
* Individuals of childbearing potential must agree to use protocol defined method(s) of contraception during the study and for at least 90-days after the last dose of IMP.
* Patients who can produce spontaneous sputum on a daily basis.
* Patients who are able to self-administer the SABA inhaler and study nebuliser for IMP administration effectively in the Investigator's opinion, following training.
* Patients appropriately vaccinated against influenza and pneumococcus at least 14-days prior to Day 1.

Exclusion Criteria:

* Currently receiving therapy with any inhaled antibiotic therapy. Patients who have previously received inhaled antibiotic therapy may be eligible if therapy was discontinued at least 28-days prior to screening.
* Treatment with systemic anti-infective therapy within 28-days prior to screening.
* Participation in other clinical studies with investigational agents within 8 weeks prior to screening.
* Treatment with NO and other NO donor agents, phosphodiesterase inhibitors and lung surfactant drugs, within 30 days prior to screening.
* Treatment with immunosuppressive medications within 2 weeks prior to screening, or systemic corticosteroids, or immunoglobulin therapy for more than 7 days within 2 weeks prior to screening.
* HIV positive AND CD4 < 350 cells/mm3
* FEV1 <55% predicted at the screening visit.
* Significant haemoptysis within 60 days of screening defined as an estimated volume of 50ml at any time.
* History of methaemoglobinaemia.
* Taking medications that may induce methaemoglobinaemia, or have received these within 30 days of screening.
* Baseline SpMet >5%.
* Current smokers of tobacco products, marijuana, e-cigarettes/vaping: a current smoker is defined as having inhaled any of these within 3 months of screening.
* In the opinion of the investigator, patients with an acute exacerbation of NCFB.
* In the opinion of the investigator, any other clinically relevant active respiratory disease with the potential to compromise participant safety or confound interpretation of safety or efficacy outcomes. Patients who have experienced >2 exacerbations of asthma or COPD requiring treatment with systemic corticosteroids within the past 12 months are not eligible.
* Asthma which requires treatment with GINA steps 4-5 suggested medications i.e., high dose ICS and LABA or leukotriene modifier/theophylline for the previous year, or systemic corticosteroids for ≥50% of the previous year to prevent it from becoming "uncontrolled", or which remains "uncontrolled" despite this therapy.
* Patients with a diagnosis of primary ciliary dyskinesia.
* Patients with a diagnosis of pulmonary hypertension.
* Patients with a current diagnosis of TB based on clinical testing or symptoms. Patients with a history of TB who have completed a course or eradication therapy at least 2 years prior to screening may be eligible if there is no clinical suspicion of recurrence. Patients with latent TB are eligible provided they have received adequate treatment per local country guidelines.
* Patients with a diagnosis, or suspected diagnosis, of NTM infection according to the ATS/IDSA statement on diagnosis, treatment, and prevention of non-tuberculous mycobacterial diseases. Patients with a previous positive culture that is suspected to be a contaminant are eligible.
* Symptomatic GERD causing NCFB disease.
* Conditions of increased risk for MetHb formation, significant anaemia or haemoglobinopathy.
* Known allergy to active substance or any excipients, or to auxiliary product.
* Known hypersensitivity to NO.
* History of anaphylaxis to any medication or hospitalisation due to an adverse drug reaction (ADR).
* Patients who are pregnant or breastfeeding.
* Patients planning to conceive a child within the anticipated period of study participation and for at least 90-days after the last dose of IMP in the study.
* Patients unable or unwilling to comply with the protocol or to cooperate fully with the investigator or site personnel.
* Alcohol or drug abuse, that in the opinion of the investigator, is sufficient to compromise the safety or cooperation of the participant.
* Patients with the following toxicities at screening as defined by the enhanced CTCAE toxicity table version 5.0, 27Nov2017.

  1. creatinine >1.5 times upper limit of normal (ULN)
  2. haemoglobin ≤8.0 g/dL
  3. platelets <50x10^9 cells/L
  4. serum potassium <3.5 mmol/L
  5. aspartate aminotransferase (AST) >3 x ULN
  6. alanine aminotransferase (ALT) >3 x ULN
  7. alkaline phosphatase (ALP) ≥ 2.5 x ULN
  8. total bilirubin >1.5 x ULN
  9. total white cell count <2 cells x 10^9/L.
* QTcF >450 milliseconds (males) or 470 milliseconds (females) or history of congenital long QT syndrome, Torsades de Pointes or other clinically significant abnormal ECG at screening or baseline.
* History of solid organ transplantation.
* History of malignancy or treatment for malignancy within the past year.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2026-02-05 (Estimated); Study Completion 2026-05-05 (Estimated)

PRIMARY OUTCOMES:
Incidence, intensity, causality, and seriousness of treatment-emergent adverse events (TEAEs). | 58 days
  A TEAE is defined as any event not present before exposure to the study treatment or any event already present that worsens in either intensity or frequency after exposure to the study treatment.
  The medical assessment of severity is determined per the CTCAE Toxicity Table Version 5 dated 27 November 2017. (Grade 1-Mild, Grade 2-Moderate, Grade 3-Severe, Grade 4 -Potentially Life threatening, Grade 5-Death)
  The relationship or association of the study treatment in causing or contributing to the AE will be characterised using the classification and criteria based on Adverse Events Attribution/Casualty Ratings Relatedness Rating table. (Not Related, Unlikely, Possible, Probable, Certain)
Changes in clinical laboratory values (haematology, clinical chemistry) at each time point. | 58 days
  The following haematological tests will be performed: haemoglobin, MetHb (local laboratory only), haematocrit, mean cell haemoglobin, mean cell volume, red blood cell count, white blood cell count with differentials (neutrophils, lymphocytes, monocytes, eosinophils, and basophils), reticulocyte count, platelet count and rheumatoid factor (Day 1 only).
  The following serum chemistry tests will be performed: albumin, blood urea nitrogen,creatinine, direct, indirect, and total bilirubin, total protein, ALP, AST, ALT, gamma-glutamyl transferase, creatinine, creatine kinase, lactate dehydrogenase, total cholesterol, calcium, sodium, potassium, chloride glucose and follicle stimulating hormone (FSH) (as required).
Changes in vital signs (blood pressure, heart rate, temperature, respiratory rate) and SpO2 at each time point. | 58 days
  Vital signs include systolic blood pressure (SBP) and diastolic blood pressure (DBP) (mmHg),heart rate (beats per minute (BPM)), respiratory rate (breaths per minute), SpO2 (%) and body temperature (axillary). On days where there is IMP dosing, vital signs should be performed prior to SABA inhaler administration and before blood draws are taken for safety assessments

SECONDARY OUTCOMES:
To characterise the PK of RESP30X in NCFB participants with confirmed high-titre respiratory PPMs. | 58 days
  Plasma PK parameter - Cmax
To characterise the PK of RESP30X in NCFB participants with confirmed high-titre respiratory PPMs. | 58 days
  Plasma PK parameter - Tmax
To characterise the PK of RESP30X in NCFB participants with confirmed high-titre respiratory PPMs. | 58 days
  Plasma PK parameter - AUC0-t,
To characterise the PK of RESP30X in NCFB participants with confirmed high-titre respiratory PPMs. | 58 days
  AUC0-tau
To characterise the PK of RESP30X in NCFB participants with confirmed high-titre respiratory PPMs. | 58 days
  Plasma PK parameter - AUC0-inf
To characterise the PK of RESP30X in NCFB participants with confirmed high-titre respiratory PPMs. | 58 days
  Plasma PK parameter - Ctrough
To characterise the PK of RESP30X in NCFB participants with confirmed high-titre respiratory PPMs. | 58 days
  Plasma PK parameter - t1/2

CONTACTS AND LOCATIONS:
Locations (1):
- ARENSIA Exploratory Medicine, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
Thirty Respiratory confirm that within one year of the end of the trial a summary of data will be uploaded to ClinTrials.gov, and all required data will be available in CTIS within the deadlines specified in relevant EU legislation. This data will remain available until the product is withdrawn from the market. This data will include but is not limited to protocol summary, safety and efficacy data related to the use of the product under the conditions of the clinical trial and which adds to the scientific understanding of the product or class of products. Patient data will be anonymised.
Time Frame: Within one year of the end of the trial, data will remain available until the product is withdrawn from the market.